CLINICAL TRIAL: NCT01333696
Title: Phase II Study of Pemetrexed Monotherapy in Patients With Platinum-resistant Squamous Cell Carcinoma of Head and Neck
Brief Title: Pemetrexed as Salvage Treatment in Squamous Cell Carcinoma of Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNTG 11-01
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Squamous cell carcinoma of head and neck; Pemetrexed
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental): 500 mg/m2, repeated every 3 weeks until disease progression or intolerable toxicity
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 at day 1. Frequence of cycles: every 3 weeks
  Other Names: Alimta

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of pemetrexed monotherapy as salvage treatment in patients with relapsed or metastatic squamous cell carcinoma of head and neck.

DETAILED DESCRIPTION:
The treatment option in patients with platinum-resistant relapsed or metastatic squamous cell carcinoma of head and neck is limited. Previous randomized phase III study showed a borderline benefit of pemetrexed added to cisplatin. Therefore, we aim to evaluate the efficacy of pemetrexed in salvage setting.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-65 years old
* Histological confirmed incurable relapsed or metastatic squamous cell carcinoma of head and neck
* Prior exposure of at least one line of platinum-containing regimen
* At least one site of measurable disease according to RECIST criteria
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Bone marrow function: ANC≧1.5×109/L, PLT≧100×109/L, Hb≧80g/L
* Liver function: total bilirubin, ALT and AST <1.5×UNL
* Renal function: Cr<1.5×UNL, CCR≧45ml/min

Exclusion Criteria:

* With curable treatment option
* Prior platinum exposure only in neo-adjuvant/adjuvant setting or concurrently used with radiotherapy
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Significant active infection
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 weeks

SECONDARY OUTCOMES:
Median progression-free survival | 1 year
Median overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China